CLINICAL TRIAL: NCT05786820
Title: Impact of a Dietary Supplementation With Maritime Pine Bark Extract (Pycnogenol®) on Gingival Inflammation - a Randomized Clinical Trial (PINEGIN)
Brief Title: Impact of Pycnogenol® on Gingival Inflammation
Acronym: PINEGIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University of Wuerzburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PINEGIN_Protocol 1.7 - 17-7-21
Record Dates: First submitted 2022-12-19; First posted 2023-03-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — pycnogenols

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled 2-arm, parallel group clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The experimental pine bark dietary supplement is packaged in neutral capsules, which are dispensed to the study patients in bottles with code labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pycnogenol Group (Active Comparator): Professional mechanical plaque removal + Pycnogenol capsule
  Interventions: Dietary Supplement: Pycnogenol
- Placebo Group (Placebo Comparator): Professional mechanical plaque removal + placebo capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pycnogenol — daily consumption of a pycnogenol-containing capsule
  Other Names: Maritime pine bark extract
  Arms: Pycnogenol Group
Dietary Supplement: Placebo — Daily consumption of a placebo capsule
  Arms: Placebo Group

SUMMARY:
This randomized, double-blind, placebo-controlled 2-arm, parallel group clinical trial is designed to evaluate the impact of the regular consumption of a polyphenol-containing Maritime Pine (Pinus pinaster) bark extract (Pycnogenol®) on clinical signs of gingival inflammation in a cohort of periodontal aftercare patients

DETAILED DESCRIPTION:
Polyphenols are natural compounds produced by plants that have various functions, such as defence against microbial pathogens or protection against UV light. Based on their antioxidant activity, a soothing or preventive effect of polyphenols on various inflammatory diseases has been suspected. There is evidence of an anti-inflammatory effect of polyphenols in manifest periodontitis as well as antibacterial properties of these compounds. In addition, it is discussed that dietary polyphenols intervene in mechanisms involved in the pathophysiology of arteriosclerotic changes and their progression.

This randomized, double-blind, placebo-controlled 2-arm, parallel group clinical trial is designed to evaluate the impact of the regular consumption of a polyphenol-containing Maritime Pine (Pinus pinaster) bark extract (Pycnogenol®) on clinical signs of gingival inflammation in a cohort of periodontal aftercare patients

ELIGIBILITY:
Inclusion Criteria:

* number of teeth ≥ 10
* age ≥ 35 ≤ 90 years
* body mass index (BMI) ≥ 20 ≤ 30
* history of periodontal disease and inclusion in a regular scheme of supportive periodontal therapy (regularly repeated subgingival biofilm removal 2-4 x/year)
* minimum of 10% probing sites displaying bleeding on probing

Exclusion Criteria:

* manifestation of inflammatory oral mucosal diseases other than gingivitis
* xerostomia (stimulated salivary flow ≤ 0.1 ml/minute)
* inability to perform regular oral home care
* inability to follow the study protocol due to intellectual or physical handicaps
* history of malignancy, radiotherapy, or chemotherapy for malignancy in the past 5 years
* current pregnancy
* acute infections such as HIV
* manifestation of metabolic bone disease
* use of antibiotics and/or anti-inflammatory medications within 4 weeks prior to screening.
* current orthodontic therapy

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing (BoP) | 6 months
  Bleeding on Probing (BoP) is defined as the appearance of a bleeding spot within 30 seconds after gently probing the evaluated periodontal pocket by inserting the periodontal probe up to the probable bottom of the pocket.

SECONDARY OUTCOMES:
Gingival Index GI | 6 months
  Gingival Index will be recorded visually according to the modification of the original GI.
Plaque Control Record (PlaCR) | 6 months
  Plaque Control Record (PlaCR) is defined as the percentage of assessed supragingival tooth surfaces covered by bacterial plaque. The presence of bacterial plaque is visually assessed after staining the tooth surfaces with a plaque staining agent.
Compositional changes within the intestinal microbiota | 6 months
  Compositional changes within the intestinal microbiota between baseline and end of the study are assessed by Next Generation Whole Genome Sequencing on a species level
Compositional changes within the oral microbiota | 6 months
  Compositional changes within the oral microbiota between baseline and end of the study are assessed by Next Generation Whole Genome Sequencing on a species level
Change in periodontally inflamed surface area (PISA) | 6 months
  PISA is calculated using the recorded pocket depths and bleeding on probing scores at each evaluated tooth at baseline and at the end of the trial at 6 months.
Change in salivary polyphenol concentration | 3 months
  Saliva samples for the analysis of salivary polyphenols levels are taken at baseline and at 3 months
Change in polyphenol serum concentration | 3 months
  Blood samples for the analysis of polyphenol serum levels are taken at baseline and at 3 months
Change in salivary levels of cytokines, cytokine inhibitors, matrix metalloproteinases and MMP inhibitors | 6 months
  Saliva samples are taken at baseline and at the end of the study at 6 months for the analysis of salivary interleukin (IL) 1ß, IL-6, IL-8, IL-31, matrix metalloproteinase (MMP)-8, MMP-9, tissue inhibitor of metalloproteinase (TIMP)-1 and Histatin 5 levels.
Change in serum levels of cytokines, cytokine inhibitors, matrix metalloproteinases and MMP inhibitors | 6 months
  Blood samples are taken at baseline and at the end of the study at 6 months for the analysis of serum interleukin (IL) 1ß, IL-6, IL-8, IL-31, matrix metalloproteinase (MMP)-8, MMP-9, and tissue inhibitor of metalloproteinase (TIMP)-1 levels.
Change in pulse wave velocity | 3 months
  Pulse wave velocity (m/sec) is measured at baseline and at 3 months
Change in central aortal pulse pressure | 3 months
  Central aortal pulse pressure (mmHg) is measured at baseline and at 3 months
Change in peripheral systolic and diastolic blood pressure | 3 months
  Peripheral systolic and diastolic blood pressure (mmHg) is measured at baseline and at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Periodontology, Center for Oral Health, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bayer J, Petersen NK, Hess JV, Jockel-Schneider Y, Hogger P. Impact of a Dietary Supplementation with French Maritime Pine Bark Extract Pycnogenol(R) on Salivary and Serum Inflammatory Biomarkers During Non-Surgical Periodontal Therapy-A Randomized Placebo-Controlled Double-Blind Trial. Nutrients. 2025 Apr 30;17(9):1546. doi: 10.3390/nu17091546. PMID 40362854